CLINICAL TRIAL: NCT05429593
Title: A Study Comparing Exposure of Semaglutide and Dapagliflozin Dosed Orally as Mono-components Versus in a Fixed-dose Combination
Brief Title: A Research Study Investigating How Semaglutide and Dapagliflozin Act in Your Body When Dosed in One Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN9917-4751; U1111-1266-4254 (Other: World Health Organization (WHO)); 2022-500007-52-00 (Other: EU CT number)
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — semaglutide; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1 sequence A (Experimental): Semaglutide followed by Semaglutide/dapagliflozin
  Interventions: Drug: Semaglutide
- Part 1 sequence B (Experimental): Semaglutide/dapagliflozin followed by Semaglutide
  Interventions: Drug: Semaglutide/dapagliflozin
- Part 2 sequence A (Experimental): Dapagliflozin followed by Semaglutide/dapagliflozin
  Interventions: Drug: Dapagliflozin
- Part 2 sequence B (Experimental): Semaglutide/dapagliflozin followed by dapagliflozin
  Interventions: Drug: Semaglutide/dapagliflozin

INTERVENTIONS:
Drug: Semaglutide — Tablet given orally
  Arms: Part 1 sequence A
Drug: Dapagliflozin — Tablet given orally
  Arms: Part 2 sequence A
Drug: Semaglutide/dapagliflozin — Tablet given orally
  Arms: Part 1 sequence B; Part 2 sequence B

SUMMARY:
This study will test how the active substances semaglutide and dapagliflozin act in the body (in terms of their levels in the blood), when they are taken in the form of a combination preparation (a tablet with a fixed dose combination) compared to when oral semaglutide and dapagliflozin are given alone.The study will consist of 2 parts. Part 1 will compare semaglutide to the fixed dose combination tablet (semaglutide/dapagliflozin) and part 2 will compare dapagliflozin to the fixed dose combination tablet (semaglutide/dapagliflozin). Participants will take part in either part 1 or part 2.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18-64 years (both inclusive) at the time of signing informed consent.
* Body mass index between 20.0 and 29.9 kg/m^2 (both inclusive).
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Participation (i.e., signed informed consent) in any other interventional, clinical study within 30 days (or 5 half-lifes of the investigational medicinal product, whichever is longer) before randomisation.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using highly-effective contraceptive method.
* Any disorder which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Use of tobacco and nicotine products, defined as any of the below:

  * Smoking more than 5 cigarettes or the equivalent per day
  * Not willing to refrain from smoking and use of nicotine substitute products during the in-house periods
* Blood donation, plasma donation or blood draw, defined as any of the below:

  * In excess of 400 mL within the past 90 days prior to the day of screening
  * In excess of 50 mL within the past 30 days prior to the day of screening
* History of major surgical procedures involving the stomach potentially affecting absorption of trial products (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery) or current presence of gastrointestinal implant.
* Presence of clinically significant gastrointestinal disorders or symptoms of gastrointestinal disorders potentially affecting absorption of drugs and/or nutrients, as judged by the investigator.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
AUC0-24h,sema,ss: area under the semaglutide plasma concentration-time curve during a dosing interval (0 to 24 hours) at steady state | From 0 to 24 hours on day 49 and 84 in Part 1
  measured in h*nmol/L
AUC0-24h,dapa,ss: area under the dapagliflozin plasma concentration-time curve during a dosing interval (0 to 24 hours) at steady state | From 0 to 24 hours on day 49 and 98 in Part 2
  measured inh*ng/mL

SECONDARY OUTCOMES:
Cmax,sema,ss: maximum observed semaglutide plasma concentration during a dosing interval (0 to 24 hours) at steady state) | From 0 to 24 hours on day 49 and 84 in Part 1
  measured in nmol/L
Cmax,dapa,ss: maximum observed dapagliflozin plasma concentration during a dosing interval (0 to 24 hours) at steady state | From 0 to 24 hours on day 49 and 98 in Part 2
  measured in ng/mL
tmax,sema,ss: time to maximum observed semaglutide plasma concentration during a dosing interval (0 to 24) at steady state | From 0 to 24 hours on day 49 and 84 in Part 1
  measured in hours
tmax,dapa,ss: time to maximum observed dapagliflozin plasma concentration during a dosing interval (0 to 24 hours) at steady state | From 0 to 24 hours on day 49 and 98 in Part 2
  measured in hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (2):
- Germany (2):
  - Novo Nordisk Investigational Site, Berlin, Brandenburg
  - Parexel International GmbH, Berlin

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com